CLINICAL TRIAL: NCT00500838
Title: CRT-D Based Impedance Monitoring Feasibility Study
Brief Title: Cardiac Resynchronization Therapy Defibrillator Based Impedance Monitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 40004384
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
Keywords: Cardiac Resynchronization Therapy; Transthoracic Impedance
MeSH Terms: conditions — Heart Failure | interventions — Cardiography, Impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- 1 (Experimental): Transthoracic impedance device implanted.
  Interventions: Device: Transthoracic Impedance

INTERVENTIONS:
Device: Transthoracic Impedance — Impedance measures will be automatically collected via the device

SUMMARY:
The intent of this feasibility study is to collect and analyze intra-thoracic impedance measurements from a CRT-D device in a heart failure population.

DETAILED DESCRIPTION:
This is a multi-center feasibility study intended to collect information on changes in intra-thoracic impedance measurements from CRT-D devices. In order to obtain an intra-thoracic impedance measurement, the device delivers a subthreshold impulse that measures the resistance between two electrodes.

At the programmed interval, measurements will be obtained between six different lead configurations.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will meet all of the following:

1. Have an approved indication per American College of Cardiology/American Heart Association/Heart Rhythm Society guidelines for implantation of a Cardiac Resynchronization Therapy Defibrillator (CRT-D) or have a previously implanted St. Jude Medical (SJM) CRT-D system capable of enabling the diagnostic impedance monitoring feature with implant occurring within the last 14 days
2. Have had at least one hospitalization, emergency department visit, or clinic visit within the past 12 months for treatment of decompensated heart failure requiring intravenous diuretics, intravenous inotropes, Natrecor (Nesiritide) therapy, or an increase in an oral diuretic of ≥100% over a 24 hour period
3. Have the ability to maintain a patient diary for recording daily weights, symptoms related to heart failure, changes in diuretic therapy, and any unscheduled clinic or hospital visits
4. Have the ability to provide informed consent for study participation and be willing and able to comply with the prescribed follow-up tests and schedule of evaluation

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

1. Be less than 18 years of age
2. Have had a recent myocardial infarction, unstable angina or cardiac revascularization within 40 days of enrollment
3. Have had a recent Cerebrovascular Accident or Transient Ischemic Attack within three months of enrollment
4. Have a contraindication for an emergency thoracotomy
5. Have an indication that requires programming device in atrial pacing mode
6. Have permanent (chronic) atrial fibrillation
7. Have a capped or inactive right atrial or right ventricular pacing/defibrillator lead
8. Have a hypersensitivity to a single 1.0mg dose of dexamethasone sodium phosphate or short term contact with heparin
9. Be pregnant or planning a pregnancy in the next 6-months
10. Be currently participating in a clinical investigation that includes an active treatment arm
11. Have a life expectancy of less than six months due to any condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the use of the impedance feature in conjunction with other functions of the CRT-D device | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: G. Stephen Greer, MD, Principal Investigator — Baptist Health
Locations (4):
- United States (4):
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Glendale Memorial Hospital, Glendale, California
  - Deborah Heart and Lung, Browns Mills, New Jersey
  - Medical University of South Carolina, Charleston, South Carolina